CLINICAL TRIAL: NCT01029002
Title: The Effects of Vitamin D Repletion in Vitamin D Deficient Patients With Stage 3 and 4 Chronic Kidney Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Albert Einstein College of Medicine (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2007-266; K23DK078774 (NIH)
Record Dates: First submitted 2009-12-07; First posted 2009-12-09 (Estimated); Results first posted 2023-08-16 (Actual); Last update posted 2023-08-16 (Actual); Status verified 2023-08

CONDITIONS: Chronic Renal Insufficiency; Proteinuria
Keywords: Vitamin D; CKD; proteinuria
MeSH Terms: conditions — Renal Insufficiency, Chronic; Proteinuria | interventions — Vitamin D

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vitamin D 50000 IU (Experimental): Patients randomized to this arm will receive 50,000 IU of ergocalciferol in one unmarked pill once weekly.
  Interventions: Drug: Vitamin D
- Placebo (Placebo Comparator): Patients randomized to this arm will receive a placebo pill once weekly.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Vitamin D — Vitamin D, ergocalciferol, 50000 IU, weekly for 12 weeks, with open label extension for another 3 months
  Arms: Vitamin D 50000 IU
Other: Placebo — Patients randomized to this arm will receive one placebo pill once weekly.
  Arms: Placebo

SUMMARY:
A randomized clinical trial to determine if vitamin D repletion in CKD (Chronic Kidney Disease) patients with low vitamin D levels will decrease proteinuria, a marker of kidney damage.

DETAILED DESCRIPTION:
This RCT will enroll 74 subjects, men and women over age of 18, with stage 3-4 CKD from various causes including diabetes and hypertension. Patients will be recruited from the Montefiore Medical Center Nephrology clinics and the Montefiore Medical Center internal medicine clinics and other interested individuals.

Informed consent will be obtained on all subjects. All subjects with meet with one of the investigators who will verbally explain to them the purpose of the study and the alternatives.

Blood and urine tests will be collected to assess for proteinuria, vitamin D levels, serum creatinine, calcium and phosphorus, as well as a urine albumin, calcium and creatinine. These tests will be used for experimental purposes only and will be collected at each study visit over the span of 6 months.

There will be two arms, an arm randomized to 50000IU of ergocalciferol once weekly and a placebo arm for 3 months. For an additional 3 months, all patients will be repleted with Vitamin D via open-label extension, based on their levels after 3 months.

Secondary outcomes include ambulatory blood pressure monitoring, hemoglobin A1c, HOMA-IR.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Ability to provide informed consent
* Chronic kidney disease stage 3 and 4
* On ACE inhibitor or ARB for albuminuria if tolerated
* Assessed during eligibility screen:
* Albuminuria >30 mg/g creatinine
* 25(OH) vitamin D level >12.5 and <75 nmol/L

Exclusion Criteria:

* On vitamin D in past 4 weeks
* Plans to relocate out of New York City in the next 6 months
* 25 (OH) Vitamin D level <12.5 nmol/L
* HIV infection
* History of hypercalcemia or kidney stones
* Serum phosphate >5.5 mg/dl in past 3 months
* Serum calcium >10.0 mg/dl in past 3 months
* SBP >160 DBP >100 at screening visit
* Transplanted organ
* Cancer
* Polycystic kidney disease
* Rapidly deteriorating kidney function with the expectation for initiation of dialysis in less than 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2009-10; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michal Melamed, MD, MHS, Principal Investigator — Albert Einstein College of Medicine
Locations (1):
- Montefiore medical center, The Bronx, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Vitamin D 50000 IU | Placebo
Started | 36 | 38
Completed | 34 | 34
Not Completed | 2 | 4
Not completed — Lost to Follow-up | 2 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vitamin D 50000 IU | Placebo | Total
Number analyzed (Participants) | 36 | 38 | 74
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.6 (9.9) | 55.3 (14.3) | 57.9 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 14 | 32
  Male | 18 | 24 | 42
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Non-Hispanic White | 3 | 3 | 6
  Non-Hispanic Black | 13 | 15 | 28
  Hispanic | 17 | 19 | 36
  Other | 3 | 1 | 4
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 36 | 38 | 74

OUTCOME MEASURES:

1. Primary Outcome: Effect of Vitamin D Supplementation on Albuminuria in CKD Patients as Assessed by Urine Albumin/Creatinine Measures.
Description: Urine albumin and creatinine were measured on spot urine specimens.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: mg/gram creatinine
Arm/Group | Vitamin D 50000 IU | Placebo
Number analyzed (Participants) | 34 | 34
mg/gram creatinine | 1126.68 (1505.26) | 1061.39 (1354.71)

2. Secondary Outcome: Effect of Repletion Doses of Vitamin D Increase 25(OH) Vitamin D Levels to Above 30 ng/mL in a Multi-ethnic Sample of Patients With CKD as a Secondary Outcome.
Description: 25(OH) vitamin D levels were measured using liquid chromatography.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Vitamin D 50000 IU | Placebo
Number analyzed (Participants) | 36 | 38
ng/mL | 29.9 (13.8) | 17.1 (7.9)

3. Secondary Outcome: Effect of Vitamin D Supplementation on Mean Systolic Blood Pressure as Measured by Ambulatory Blood Pressure in CKD Patients as a Secondary Outcome.
Time Frame: 3 months
Population: Ambulatory pressure data readings were not collected and therefore data was not able to be aggregated and analyzed.
Arm/Group | Vitamin D 50000 IU | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Vitamin D 50000 IU | Placebo
All-Cause Mortality (participants affected / at risk) | 0/36 | 0/38
Serious Adverse Events (participants affected / at risk) | 12/36 | 17/38
Other Adverse Events (participants affected / at risk) | 0/36 | 0/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vitamin D 50000 IU (N=36) | Placebo (N=38)
Cardiac Hospitalization and ED Visits (Cardiac disorders) | 3 (3) | 6 (6)
Non-cardiac Hospitalization and ED Visits (General disorders) | 9 | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes